CLINICAL TRIAL: NCT00272935
Title: A Randomized, Multicenter, Double-blind, Placebo-controlled Trial to Demonstrate the Safety and Efficacy of Daily 0.3 mg Synthetic Conjugated Estrogens, A (Cenestin) for the Treatment of Vasomotor Symptoms in Postmenopausal Women
Brief Title: A Clinical Trial to Demonstrate the Efficacy and Safety of Cenestin 0.3 mg for the Treatment of Hot Flashes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Duramed Protocol Chair, Duramed Research, Inc.
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BR-CEN-301
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2009-07

CONDITIONS: Hot Flashes
Keywords: menopause; vasomotor symptoms
MeSH Terms: conditions — Hot Flashes | interventions — estrogens, conjugated synthetic A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Cenestin 0.3 mg Tablets
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cenestin 0.3 mg Tablets — 1 tablet daily
  Other Names: Synthetic conjugated estrogens, A
  Arms: 1
Other: Placebo — 1 tablet daily
  Other Names: Placebo tablets
  Arms: 2

SUMMARY:
This is a randomized, double-blind study to compare the efficacy and safety of daily doses of Cenestin 0.3 mg tablets to placebo in reducing the frequency and severity of moderate to severe hot flashes in postmenopausal women.

DETAILED DESCRIPTION:
The overall study duration will be approximately 16 weeks. After a screening/baseline period of up to 4 weeks patients will be randomized to receive either placebo tablets or Cenestin 0.3mg tablets

ELIGIBILITY:
Inclusion Criteria:

* Naturally or surgically postmenopausal
* At least 12 months since last menses or 6 weeks past surgery
* Minimum of 7 daily or 50 weekly moderate to severe hot flashes

Exclusion Criteria:

* Any contraindication to natural or synthetic estrogens

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Mean change in average frequency of moderate to severe hot flashes | Baseline to Day 28 and to Day 84
Mean change in severity of moderate to severe hot flashes | Baseline to Day 28 and to Day 84

SECONDARY OUTCOMES:
Safety and tolerability of Cenestin 0.3mg | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Research Protocol Chair, Study Chair — Duramed Research, Inc
Locations (43):
- United States (43):
  - Duramed Investigational Site, Huntsville, Alabama
  - Duramed Investigational Site, Montgomery, Alabama
  - Duramed Investigational Site, Phoenix, Arizona
  - Duramed Investigational Site, Tucson, Arizona
  - Duramed Investigational Site, Carmichael, California
  - Duramed Investigational Site, Irvine, California
  - Duramed Investigational Site, San Diego, California
  - Duramed Investigational Site, San Ramon, California
  - Duramed Investigational Site, Brooksville, Florida
  - Duramed Investigational Site, Coral Gables, Florida
  - Duramed Investigational Site, Gainesville, Florida
  - Duramed Investigational Site, Leesburg, Florida
  - Duramed Investigational Site, Miami, Florida
  - Duramed Investigational Site, Palm Springs, Florida
  - Duramed Investigational Site, Venice, Florida
  - Duramed Investigational Site, Alpharetta, Georgia
  - Duramed Investigational Site, Douglasville, Georgia
  - Duramed Investigational Site, Boise, Idaho
  - Duramed Investigational Site, Evansville, Indiana
  - Duramed Investigational Site, Lexington, Kentucky
  - Duramed Investigational Site, Baltimore, Maryland
  - Duramed Investigational Site, Lincoln, Nebraska
  - Duramed Investigational Site, Las Vegas, Nevada
  - Duramed Investigational Site, Albuquerque, New Mexico
  - Duramed Investigational Site, Cleveland, Ohio
  - Duramed Investigational Site, Columbus, Ohio
  - Duramed Investigational Site, Mayfield Heights, Ohio
  - Duramed Investigational Site, Medford, Oregon
  - Duramed Investigational Site, King of Prussia, Pennsylvania
  - Duramed Investigational Site, North Wales, Pennsylvania
  - Duramed Investigational Site, Philadelphia, Pennsylvania
  - Duramed Investigational Site, Pittsburgh, Pennsylvania
  - Duramed Investigational Site, Charleston, South Carolina
  - Duramed Investigational Site, Bristol, Tennessee
  - Duramed Investigational Site, Clarksville, Tennessee
  - Duramed Investigational Site, Nashville, Tennessee
  - Duramed Investigational Site, Dallas, Texas
  - Duramed Investigational Site, Fort Worth, Texas
  - Duramed Investigational Site, Houston, Texas
  - Duramed Investigational Site, San Antonio, Texas
  - Duramed Investigational Site, Norfolk, Virginia
  - Duramed Investigational Site, Spokane, Washington
  - Duramed Investigational Site, Tacoma, Washington